CLINICAL TRIAL: NCT02867540
Title: Comparison of Endoscopy and Diffusion-weighted Enterography-MRI for the Diagnosis of Crohn's Disease Recurrence Following Ileocolic Resection: a Pilot Study
Acronym: MRI-CROHN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA14058
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

ARMS (1):
- experimental group (Experimental): Patient's with Crohn's disease who have had ileocolic resection
  Interventions: Other: MRI enterography

INTERVENTIONS:
Other: MRI enterography

SUMMARY:
Nearly three-quarters of patients with Crohn's disease have small bowel involvement and 80% of them will have complications that will require a surgical procedure, usually an ileocolonic resection with ileocolonic anastomosis. The rate of recurrence at the anastomosis site and in the ileum after surgery, whether symptomatic or not, is high, at least 60% in one year and 80% within three years. The gold standard for monitoring being ileocolonoscopy, endoscopic surveillance is recommended in these patients, once between 6 to 12 months after surgery and then every 2 years.

The MRI enterography is a validated technique for the assessment of small bowel Crohn's disease. The enterography MRI is a validated technique for the assessment of small bowel Crohn's disease. The MRI enteroclysis was evaluated in two studies compared to endoscopy, with excellent performance in terms of recurrence detection sensitivity and suggested as an alternative to it to avoid an invasive procedure repeated in these patients. The MRI enterography (without enteroclysis) does not provide as good distension of the bowel loops as MRI enteroclysis because it relies on the principle of oral ingestion prior to the examination of large amounts of liquid. However, it is much better tolerated by the patient, does not involve radiation that exists with enteroclysis, is much simpler to use and requires no special equipment to magnetic fields.

DETAILED DESCRIPTION:
Determine the diagnostic performances of MRI enterography for the diagnosis of recurrence at the anastomosis site and in the ileum in patients with Crohn's disease who have had ileocolonic resection.

Assess the value of diffusion sequences of MRI enterography for the diagnosis of recurrence at the anastomosis site and in the ileum in patients with Crohn's disease who have had ileocolonic resection.

ELIGIBILITY:
Inclusion Criteria:

* patients with Crohn's disease
* patients with ileocolonic resection more than 6 months ago and less than 4 years ago
* patients with indication of ileocolonoscopy
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

* patients with contraindications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
recurrence at the anastomosis site and in the ileum | Day 1
  Recurrence diagnosed with colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France